CLINICAL TRIAL: NCT04917952
Title: Effectiveness of Blood Flow Restriction (BFR) Exercise Therapy to Reduce Pain in Knee Osteoarthritis (OA) Patients. A Double-blinded Randomised Clinical Trial
Brief Title: Effectiveness of Blood Flow Restriction Exercise Therapy to Reduce Pain in Knee Osteoarthritis Patients
Acronym: BFR;OA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of West Attica (Other)
Responsible Party: Principal Investigator, Christos Anagnostis, Principal Investigator, University of West Attica
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 36676 - 27/04/202
Record Dates: First submitted 2021-05-25; First posted 2021-06-08 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Knee Osteoarthritis
Keywords: chronic pain
MeSH Terms: conditions — Osteoarthritis, Knee; Chronic Pain | interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- BFR group (Experimental): The intervention group will receive resisted knee extension 30% of 1RM with blood flow restriction.
  Interventions: Device: Blood Flow Restriction (BFR)
- Sham BFR group (Placebo Comparator): The control group will receive resisted knee extension 30% of 1RM with sham blood flow restriction.
  Interventions: Device: Sham Blood Flow Restriction (sham BFR)

INTERVENTIONS:
Device: Blood Flow Restriction (BFR) — * Exercise: Bilateral knee extension at range 90ο-0ο
  * Load: 30% 1RM
  * BFR: Yes, 80% at both legs
  * Sets: 4
  * Reps: 30-15-15-15
  * Rest: 30'' between sets
  * Tempo: 2-0-2-0
  Participants of the intervention group will receive an exercise protocol with blood flow restriction once and will be measured for changes in PPT by the use of a digital dynamometer.
  Exercise protocol will be four sets of bilateral knee extension 90ο-0ο, reps per set 30-15-15-15, tempo 2-0-2-0 and rest 30 sec between sets.
  In order to determine the training load 30% of 1RM, participants will perform bilateral knee extension in range 90ο-0ο with pain-free maximum resistance. The derived 1RM will be used to determine the 30% 1RM load.
  Blood flow restriction will be applied at 80% by using pressure cuffs. The cuffs will be applied to the proximal thigh. Cuff pressure needed for a 100% vascular occlusion will be determined for each individual at a seated and relaxed position.
  Other Names: Kaatsu
  Arms: BFR group
Device: Sham Blood Flow Restriction (sham BFR) — * Exercise: Bilateral knee extension at range 90ο-0ο
  * Load: 30% 1RM
  * BFR: Yes, Sham BFR, 10mm Hg at both legs
  * Sets: 4
  * Reps: 30-15-15-15
  * Rest: 30'' between sets
  * Tempo: 2-0-2-0
  Participants of the control group will receive an exercise protocol with sham blood flow restriction once and will be measured for changes in PPT by the use of a digital dynamometer.
  Exercise protocol will be four sets of bilateral knee extension 90ο-0ο, reps per set 30-15-15-15, tempo 2-0-2-0 and rest 30 sec between sets.
  In order to determine the training load 30% of 1RM, participants will perform bilateral knee extension in range 90ο-0ο with pain-free maximum resistance. The derived 1RM will be used to determine the 30% 1RM load.
  Sham technique for blood flow restriction will be applied by using pressure cuffs inflated at 10mm Hg. The cuffs will be applied to the proximal thigh. Cuff pressure will be applied for each individual at a seated and relaxed position.
  Other Names: Sham Kaatsu
  Arms: Sham BFR group

SUMMARY:
Resistance training of knee extensor muscles is being used in physiotherapy management in knee osteoarthritis (OA) to improve pain and physical function. Blood flow restriction (BFR) has been suggested to improve pain and increase muscle strength in healthy subjects and certain diseases. Although there are clinical studies suggesting improvements in knee osteoarthritis symptoms after 4-12 weeks of exercise with BFR, the acute effects of the intervention have not been known.

This study aims to assess the effectiveness of low load exercise therapy combined with BFR on acute pain reduction and within 24 hours post-intervention on people with knee OA compared to a placebo group.

This study will take place in Athens, Greece, as part of the postgraduate MSc program of the Physiotherapy department of the University of West Attica.

DETAILED DESCRIPTION:
A double-blinded randomised clinical trial with a total of 42 participants will be randomly assigned to the intervention (n=21) or the control group (n=21).

The intervention group will complete a single exercise session with BFR 80%, 30% 1RM, while the control group will have sham BFR, 30% 1RM.

Pain Pressure Threshold (PPT) will be assessed with the use of a digital pressure dynamometer.

ELIGIBILITY:
Inclusion Criteria:

* Current osteoarthritis clinical diagnosis according to either European League Against Rheumatism (EULAR) or American College of Rheumatology (ACR) criteria
* VAS/NRS Knee pain ≥3/10 during activity

Exclusion Criteria:

* Previous experience with BFR
* Has followed knee exercise or kinesiotherapy program in the past 3 months
* New medicines in the past 3 months
* Any lower limb surgery in the past 6 months
* Knee arthroplasty surgery (Knee replacement)
* Any active healing process affecting walking (fracture, sprain, strain, etc.)
* Diagnosed with rheumatologic/neurologic disease affecting functionality
* Diagnosed or history of heart or vascular diseases
* Diagnosed with respiratory/metabolic disease
* Personal history of cancer
* Cognitive problems
* Pregnancy (only for female participants)
* Any other indication not to participate in exercise

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Change of Pain Pressure Threshold (PPT) from baseline | At baseline, Post 5 minutes, Post 24 hours
  Pain will be measured with a digital dynamometer. Raise of the PPT value means a better outcome

SECONDARY OUTCOMES:
Change of Dynamic weight-bearing Assessment of Pain (DAP) from baseline | At baseline, Post 5 minutes, Post 24 hours
  DAP is correlating VAS/NRS pain reporting scales with the functional test of 30-second Chair Stand Test (30s-CST)
Change of 30-second Chair Stand Test (30s-CST) from baseline | At baseline, Post 5 minutes, Post 24 hours
  30s-CST is a functional assessment evaluating leg strength and dynamic balance, the more repetitions one can do during the 30'', the better the outcome
Change of pain score from baseline with the use of reporting scales Visual Analogue Scale (VAS) / Numeric Rating Scale (NRS) | At baseline, Post 5 minutes, Post 24 hours
  Pain reporting scales as NRS are using 0-10 grades to measure how big the pain is, 10 is for the worst pain

OTHER OUTCOMES:
Douleur Neuropathique 4 questionnaire (DN4 greek) | At least 72 hours prior the intervention
  Greek version of DN4 will be used diagnostically to identify the existence of neuropathic pain, a score greater than 4/10 suggests the existence of neuropathic pain
Knee Osteoarthritis Outcome Scale (KOOS greek) | At least 72 hours prior the intervention
  Greek version of the KOOS will be used diagnostically to identify the severity of the disease. Each category score ranges 0-100, the minimum score is the worst
1 Repetition Maximum (1RM) | At least 72 hours prior the intervention
  1RM will be used diagnostically to identify the maximum strength of the participants. Each participant will extend their knees bilaterally, pain-free, 90o-0ο with the maximum weight
Other demographics and medical notes | At least 72 hours prior the intervention
  Recording of demographics and medical notes will be used to identify the inclusion and exclusion criteria

CONTACTS AND LOCATIONS:
Overall Officials: George Gioftsos, Study Director — University of West Attica

IPD SHARING:
Plan to Share IPD: No